CLINICAL TRIAL: NCT07144124
Title: The Effect of Probiotic Supplementation on the Incidence of ICU-Acquired Infections Among Enterally Fed Patients: A Single-Center, Randomized, Open-Label, Controlled Pilot Trial
Brief Title: Probiotics for Preventing ICU-Acquired Infections in Critically Ill Patients: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Aqdar Mufareh Al Aklabi, Principal Investigator, Master's Candidate in Clinical Nutrition, and Clinical Dietitian at Almana Medical Center - Rakah, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-77
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cross Infection (Hospital-Acquired Infections); Critical Illness; Probiotic Intervention
MeSH Terms: conditions — Cross Infection; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1: Control Group - Standard ICU Care (No Intervention): Participants in this arm will receive standard ICU care according to institutional protocols. No probiotic supplementation will be administered.
- Probiotic Group - Standard Care Plus Biopro-Max (Experimental): Participants in this arm will receive standard ICU care according to institutional protocols plus Biopro-Max 8 Billion Probiotics (Bioserv Healthcare). The supplement will be administered as one bottle per day for 15 consecutive days.
  Interventions: Dietary Supplement: Biopro-max 8 Billion Probiotics (Bioserv Healthcare)

INTERVENTIONS:
Dietary Supplement: Biopro-max 8 Billion Probiotics (Bioserv Healthcare) — Participants in the intervention arm will receive Biopro-Max 8 Billion Probiotics (Bioserv Healthcare). The supplement will be administered as one bottle per day for 15 consecutive days in addition to standard ICU care. The intervention is intended to evaluate whether daily probiotic supplementation reduces the incidence of ICU-acquired infections and improves related clinical outcomes, including inflammatory and immune markers, feeding tolerance, muscle changes, and mortality.
  Arms: Probiotic Group - Standard Care Plus Biopro-Max

SUMMARY:
This pilot randomized clinical trial investigated the effect of probiotic supplementation on the incidence of intensive care unit-acquired infections (ICU-AIs) in critically ill patients. ICU-AIs are a major complication in patients receiving mechanical ventilation and enteral nutrition, contributing to increased morbidity, prolonged ICU length of stay, and higher mortality rates.

The objective of this study was to assess whether daily administration of a probiotic supplement, in addition to standard ICU care, could reduce the risk of ICU-AIs compared with standard care alone. Eligible participants were critically ill adults who were mechanically ventilated and receiving enteral feeding. Patients were randomly assigned to one of two groups:

Control group: standard ICU care. Intervention group: standard ICU care plus probiotic supplementation (Biopro-max 8 Billion Probiotics (Bioserv Healthcare)).

The intervention continued for 15 days, during which participants were monitored daily for the occurrence of ICU-AIs confirmed by the treating ICU physician. Secondary outcomes included inflammatory and immune markers (CRP, PCT, IgG, IgA), tolerance to enteral feeding, skeletal muscle changes assessed by point-of-care ultrasound, ICU and hospital length of stay, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled patients were critically ill adults aged 18 years or older, had initiated enteral nutrition (EN) within 48 hours of ICU admission, were required mechanical ventilation and were anticipated to remain ventilated for at least five days.

Exclusion Criteria:

* Patients were excluded if they had been mechanically ventilated for more than 72 hours before enrollment; had an absolute neutrophil count under 500/mm³; had received antibiotics for more than three days before screening; had received immunosuppressants within one week prior to enrollment or had a diagnosis of immunosuppressive disease; had end-stage cancer; had previously received probiotics, prebiotics, or synbiotics before screening; were pregnant or lactating; or had not received the first dose of probiotics within 48 hours following ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
Incidence of ICU-Acquired Infections. | Within 15 days from enrollment or until ICU discharge, whichever occurs first.
  ICU-acquired infections are defined as infections that were not present or detected at ICU admission but occurred during the ICU stay. Infections were confirmed by the attending ICU physician.

SECONDARY OUTCOMES:
Inflammatory Marker Levels (CRP and PCT) | Baseline, Day 5, Day 10, and Day 15
  Monitor changes in serum CRP and PCT levels at different timepoints to evaluate systemic inflammation.
Immunoglobulin Levels (IgG and IgA) | Baseline, Day 5, Day 10, and Day 15
  Monitor changes in serum IgG and IgA levels at different timepoints to assess immune function.
Enteral Feeding Intolerance | Daily for 15 days or until ICU discharge
  Monitor the occurrence of enteral feeding intolerance based on gastric residual volume, abdominal distention, vomiting, diarrhea, and use of prokinetic drugs.
Muscle wasting | Baseline, Day 5, Day 10, and Day 15
  Monitor changes in rectus femoris and vastus intermedius muscle thickness using ultrasound at different timepoint
Mortality | Within 15 days after enrollment.
  Monitor the number of deaths that occur during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- King Fahad Military Medical Complex, Dhahran, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the small sample size and privacy concerns.